CLINICAL TRIAL: NCT06820476
Title: Investigation of Safety, Tolerability and Pharmacokinetic Properties of Multiple Oral Doses of NNC0487-0111 in Chinese Participants With Overweight or Obesity
Brief Title: A Research Study on How NNC0487-0111, a New Medicine, Works in Chinese Participants After 10 Days of Oral Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9487-7573; U1111-1289-3164 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NNC0487-0111 (dose 1) (Experimental): Participants will be randomized to receive a single dose of NNC0487-0111.
  Interventions: Drug: NNC0487-0111
- NNC0487-0111 (dose 2) (Experimental): Participants will be randomized to receive a single dose of NNC0487-0111.
  Interventions: Drug: NNC0487-0111
- NNC0487-0111 (dose 3) (Experimental): Participants will be randomized to receive a single dose of NNC0487-0111.
  Interventions: Drug: NNC0487-0111
- Placebo (Placebo Comparator): Participants will be randomized to receive matching Placebo to NNC0487-0111.
  Interventions: Drug: Placebo (NNC0487-0111)

INTERVENTIONS:
Drug: NNC0487-0111 — Participants will be randomized to receive NNC0487-0111 tablet orally at dose levels 1, 2, or 3.
  Arms: NNC0487-0111 (dose 1); NNC0487-0111 (dose 2); NNC0487-0111 (dose 3)
Drug: Placebo (NNC0487-0111) — Participants will be randomized to receive a placebo tablet orally matched to NNC0487-0111.
  Arms: Placebo

SUMMARY:
The study is testing a new study medicine called NNC0487-0111 for weight control in Chinese people with Body mass index (BMI) greater than or equal to (>=) 24 kilogram per square meter (kg/m^2). The aim of this study is to find out how safe the study medicine is and how it behaves in your body. Participants will either get NNC0487-0111 or placebo. Which treatment participants will get is decided by chance. Oral NNC0487-0111 is a new medicine which cannot be prescribed by doctors but has previously been tested in humans. The study will last for about 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male Chinese participants, age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 24.0 and 34.9 kilogram per square meter (kg/m^2)(both inclusive), with a body weight greater than or equal to (>=) 65.0 kilogram (kg), at screening.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder, unwillingness or inability which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Glycated haemoglobin (HbA1c) greater than or equal to (>=) 6.5 percent (%) (48 millimoles per mole [mmol/mol]) at screening
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values:
* Vitamin D (25-hydroxycholecalciferol) less than (<) 12 Nanograms per millilitre (ng/mL) (30 nanometer[nM]) at screening
* Parathyroid hormone (PTH) outside normal range at screening
* Total calcium outside normal range at screening
* Amylase greater than or equal to (>=) 2 times upper limit of normal at screening
* Lipase greater than or equal to (>=) 2 times upper limit of normal at screening
* Calcitonin greater than or equal to (>=) 50 picograms per milliliter (pg/mL) at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2025-02-09 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From first NNC0487-0111 administration (Day 1) to completion of the end-of-study visit (Day 31)
  Number of events

SECONDARY OUTCOMES:
AUC0-24h,MD; the area under the NNC0487-0111 plasma concentration-time curve from time 0 to 24 hours after last multiple dose | From pre-dose on Day 10 until Day 11
  measured in hour*nanomoles per liter (h*nmol/L)
Cmax,MD; the maximum plasma concentration of NNC0487-0111 after last multiple dose | From pre-dose on Day 10 to completion of the end-of-study visit (Day 31)
  measured in nanomoles per liter(nmol/L)
tmax,MD; the time of maximum plasma concentration of NNC0487-0111 after last multiple dose | From pre-dose on Day 10 to completion of the end-of-study visit (Day 31)
  measured in hour (h)
Change in bodyweight | From baseline Day 1 to Day 11
  measured in percentage (%)
Change in fasting plasma glucose | From baseline Day 1 to Day 11
  measured in millimoles per liter (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- China (2):
  - Jinan Central Hospital Affiliated to Shandong University, Ji'Nan, Shandong
  - Jinan Central Hospital, Ji'Nan, Shandong

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com